CLINICAL TRIAL: NCT06553170
Title: Anesthetic Management of Diabetes in Perioperative Urology and Visceral Surgery: Adherence to a New Protocol at Brest CHU
Brief Title: Anesthetic Management of Diabetes in Perioperative Urology and Visceral Surgery
Acronym: DIAPRO-BREST
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DIAPRO-BREST (29BRC18.0128)
Record Dates: First submitted 2021-06-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; glycemic balance; anesthesia; perioperative medecine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before: all patients before the presentation of new protocol about management of diabètes in perioperative urology et visceral surgery
- after: all patients after the presentation of new protocol about management of diabètes in perioperative urology et visceral surgery

SUMMARY:
It is recognized that a poor glycemic, pre- and intraoperative balance is the source of increase in morbimortality. There was no local protocol at the CHRU Brest regarding the perioperative management of the diabetic patient. This retrospective observational work aims to assess the application of the French recommendations for the perioperative management of diabetes, and compare management before and after the introduction of a protocol based on its recommendations published in 2017 by the SFAR.

The main endpoint is the percentage of patients for whom half of the patients recommendations from the local protocol were implemented for each of the recommendations evaluated and applicable to each patient, before and after protocol and staff training.

DETAILED DESCRIPTION:
Half of the recommandations are implemented for each recommendation evaluated applicable in 29% of patients(n=25) in the before group versus 66.23% (n=52) in the after group (p<0.05).

This corresponds to an improvement significant of 36.23% for our primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* patients diabetics
* urology or visceral surgery

Exclusion Criteria:

* ambulatory surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients diabetics in Brest CHU
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
follow the recommendations | 1 year after
  The main endpoint is the percentage of patients for whom half of patients recommendations of the local protocol were implemented for each of the recommendations evaluated and applicable to each patient, before and after the application of the protocol and training staff.

SECONDARY OUTCOMES:
complications and mortality | 1 year after
  Secondary endpoints are hospital mortality, the occurrence of early postoperative complications related to diabetes, the occurrence of complications post-operative surgery, and finally the occurrence of medical complications not related to Diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: anna cadic, Principal Investigator — chru brest, france
Locations (1):
- Cadic, Brest, Brittany Region, France